CLINICAL TRIAL: NCT01900353
Title: Vertical Versus Horizontal Brushing: a Randomized Split-mouth Clinical Trial
Brief Title: Vertical vs Horizontal Brushing: a Randomized Split-mouth Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Maria Grazia Cagetti, Assistant professor senior researcher, University of Milan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012CC01
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Dental Plaque
MeSH Terms: conditions — Dental Plaque

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- horizontal brushing method (Active Comparator): brushing methods
  Interventions: Other: brushing methods
- Vertical brushing method (Active Comparator): brushing methods
  Interventions: Other: brushing methods

INTERVENTIONS:
Other: brushing methods

SUMMARY:
The aim of this randomized, single-blind, split-mouth design, clinical trial was to evaluate the effectiveness in plaque removal of the vertical and the horizontal brushing methods. Trauma on soft tissues were also registered. Sixty-one (61) young adults were enrolled for this trial and forty-three (43) completed the brushing session. All subject were asked to abstain from oral hygiene procedures for 48 hours before the brushing session to allow adequate plaque accumulation. They were firstly instructed to use a dental disclosing tablet in order to easily permit to detect dental plaque on teeth and to highlight soft tissue abrasions. Plaque and the abrasion indexes were recorded according to the Rustogi Modified Navy Plaque Index (RMNPI) and the Danser Index (DI) by the same examiner. The brushing session was always performed by the same dental hygienist who brush with a randomized split-mouth design. After the brushing session, the blinded examiner recorded the indexes again.

DETAILED DESCRIPTION:
Study population The study was conducted from October 2012 to December 2012 in the Dental Clinic of San Paolo Hospital in Milan. Sixty-one (61) students (19-24 years) attending the Dental Clinic were contacted with an information leaflet, explaining the aim of the study and requesting their participation with signed consent. Forty-nine (80.33% of total sample) agree to participate and underwent to an oral examination. The presence of seven evaluable teeth in each quadrant was considered the inclusion criterion. Exclusion criteria were the presence of oral mucosal lesions, periodontal pocket ≥ 4 mm, gingival recession, orthodontic treatment, caries lesions in buccal and/or lingual surfaces, removable prosthesis, use of mouthrinses containing plaque-reducing agents (e.g. chlorhexidine, essential oils, cetylpyridinium chloride) on regular basis.

One (1) subject was excluded because of the presence of periodontal pockets. Forty-eight (48) young adults were enrolled, five (10.42% drop-out rate) subjects did not attend the scheduled appointment and so the study reports data on 43 subjects.

All subjects were given a thorough professional prophylaxis to remove plaque, stains and calculus. The study protocol was approved by the Ethical Committee of San Paolo Hospital.

Study design and calibration of the personnel The study was designed and performed as split-mouth design. The subjects were listed and a list of true random numbers was generated (www.random.org). The generator was set to produce a true random sequence of "1" and "2", where "1" represented a mouth in which first and third quadrants were brushed with vertical method and "2" in which second and fourth quadrants were brushed with the same method.

A dental hygienist performed the brushing sessions. A calibration course was carried out one week before the starting of the study. She applied the two brushing methods first on Columbia Dentoform® and after on 2 volunteers.

Clinical parameters were recorded by one examiner (SM), using a mouth plane mirror (Hu-Friedy, Nr. 5, diameter mm 24) and a millimeter periodontal probe (Hu-Friedy, CP-15,5B - Qulix) under optimal artificial lighting. The examiner (SM) was previously calibrated.

Toothbrushing Subjects were asked to abstain from oral hygiene procedures for 48 hours before the brushing session to allow adequate plaque accumulation. Before the brushing session, all subjects used a dental disclosing tablet (Red-Cote, D&C Red #28, 1.5% w/w, Sunstar Suisse S.A., 20147 Saronno, Italy) to easily detect dental plaque on teeth and to highlight soft tissue abrasions following strictly the manufacturer's directions: rinse mouth with water, chew a tablet swishing around for 30 seconds, expectorate, and rinse again with water.

The same model of manual toothbrush was used for all subjects (Mentadent Tecnic Clean, Medium, Unilever Austria GmbH, 1023 Wien). The number of movements of the bristles on each tooth surfaces was set as five.

In the vertical toothbrushing method, the dental hygienist placed the bristles on the gingival margin of the teeth (two teeth are generally covered by toothbrush head) and moved the toothbrush in the occlusal direction; this movement was repeated five times for each couple of teeth, for buccal and lingual side. In the horizontal toothbrushing method, the bristles were placed on the teeth surfaces (the width of the toothbrush head covered the entire tooth surface) and moved distal to mesial and mesial to distal until the fifth movement was reached. The movements were performed one for posterior teeth and one for anterior teeth (canine and lateral incisor.

At the end of the brushing session, subjects were invited to repeat the disclosing procedure to highlight soft tissue abrasions produced by the bristles.

Plaque index evaluation The plaque scores were recorded two times, before and after the brushing, by one examiner (SM). The Rustogi Modified Navy Plaque Index was used(Rustogi 1992). The index evaluates 18 records. The buccal and the lingual surfaces of each tooth are ideally divided in 9 areas, scored as 0 (absence of disclosed plaque) or 1 (presence of disclosed plaque). The 9 areas are called a, b, c, d, e, f, g, h and i and they refer to the whole buccal and lingual surfaces: areas a, b and c refer to the gingival margin, areas d and f to approximal surfaces, areas e,h, and g to the middle areas of the surface and finally, area i refers to cuspal margin.

The mean plaque scores was calculated for the whole tooth surface, the gingival and in the interproximal areas scores for each subject.

The third molars, if present, were excluded from recordings. Plaque index of the central incisors was not considered because of the over-brushing depending on the split-mouth design of the study.

Gingival abrasions evaluation Gingival abrasions were assessed utilizing the method adapted by Danser (Danser 1998). The gingival tissues were divided into three areas defined as marginal for the marginal free gingiva, interdental for the papillary-free gingiva and mid-gingival for the attached gingiva. In the upper jaw the palatal mid-gingival area comprised the whole hard palate. The abrasions were measured using a periodontal probe placed along the axis of the lesion; they were classified as small (≥ 2 mm), medium (≥ 3 mm but ≤ 5 mm) and large (> 5 mm).

ELIGIBILITY:
Inclusion Criteria:

* seven evaluable teeth in each quadrant

Exclusion Criteria:

* the presence of oral mucosal lesions, periodontal pocket ≥ 4 mm, gingival recession, orthodontic treatment, caries lesions in buccal and/or lingual surfaces, removable prosthesis, use of mouthrinses containing plaque-reducing agents (e.g. chlorhexidine, essential oils, cetylpyridinium chloride) on regular basis.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
dental plaque score | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grazia Cagetti, DDS PhD, Principal Investigator — Department of Health Sciences, University of Milan
Locations (1):
- Dental Clinic San Paolo Hospital, Milan, Italy

REFERENCES:
- [Background] Ganss C, Schlueter N, Preiss S, Klimek J. Tooth brushing habits in uninstructed adults--frequency, technique, duration and force. Clin Oral Investig. 2009 Jun;13(2):203-8. doi: 10.1007/s00784-008-0230-8. Epub 2008 Oct 14. PMID 18853203